CLINICAL TRIAL: NCT02416505
Title: The Age of OrthoInfo: A Randomized Controlled Trial Evaluating Patient Comprehension of Informed Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Nkemakolam Egekeze, Orthopedic Surgery Researcher, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-334
Record Dates: First submitted 2015-04-06; First posted 2015-04-15 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Verbal Discussion: Control Group (No Intervention): In this group, participants will receive a 10 minute Verbal Only Knee Osteoarthritis Steroid Injection Informed Consent discussion.
  This discussion will cover the relevant topics of Knee OA causes, relevant anatomy, symptoms, diagnosis, and treatment options. This discussion will also include the risks, benefits, and alternatives to a steroid injection.
- Verbal+Anatomic Model (Active Comparator): This intervention group will receive a 10 minute Knee Osteoarthritis Steroid Injection Informed Consent discussion with the aid of a Knee Model.
  This discussion will cover the relevant topics of Knee OA causes, relevant anatomy, symptoms, diagnosis, and treatment options. This discussion will also include the risks, benefits, and alternatives to a steroid injection.
  Interventions: Behavioral: Verbal+Anatomic Model
- Verbal+Video Presentation (Active Comparator): This intervention group will receive a 10 minute Knee Osteoarthritis Steroid Injection Informed Consent discussion with the aid of a Video.
  This discussion will cover the relevant topics of Knee OA causes, relevant anatomy, symptoms, diagnosis, and treatment options. This discussion will also include the risks, benefits, and alternatives to a steroid injection.
  Interventions: Behavioral: Verbal+Video

INTERVENTIONS:
Behavioral: Verbal+Anatomic Model
  Arms: Verbal+Anatomic Model
Behavioral: Verbal+Video
  Arms: Verbal+Video Presentation

SUMMARY:
This study is a Non-funded, Single Center, Multi-Arm, Parallel Group Randomize Control Trial.

In this study, the investigators aim to evaluate the impact of a visual aid on patient comprehension an orthopedic informed consent discussion in low socioeconomic populations.

The primary outcome is patient comprehension measured by a Validated Knowledge-Based Multiple Choice Questionnaire.

The secondary outcomes include: Patient satisfaction and Time efficiency.

The investigators hypothesize that using an Anatomic Model Visual Aid during an orthopedic informed consent discussion will improve patient comprehension, satisfaction and time-efficiency of orthopedic care.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with Knee Osteoarthritis managed with steroid injections
* Patients who express lack of knowledge regarding knee osteoarthritis (causes, diagnosis, treatment, anatomy)
* English speaking
* Patients that meet the Federal Poverty Guideline for Healthcare (i.e. Medicaid)

Exclusion Criteria:

* Patients under the age of 18
* College graduates
* Non-English speaking
* Patient without the capacity to give consent
* Patients with a tactile, mental, visual or auditory disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The Nkem Test | 20 minutes
  Comprehension based examination of an informed consent discussion

SECONDARY OUTCOMES:
Patient Satisfaction Survey | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bernhardt, MD, Study Chair — UMKC Department of Orthopaedic Surgery; Johnathan Dubin, MD, Study Director — UMKC Department of Orthopaedic Surgery; Karen Williams, PhD, Study Director — UMKC Dept of Bioinformatics; Nkem Egekeze, MD, Principal Investigator — UMKC Dept of Orthopaedic Surgery